CLINICAL TRIAL: NCT02166333
Title: Vitamin D Supplements to Prevent Falls in Older Adults: A Dose-Response Trial
Brief Title: Study To Understand Fall Reduction and Vitamin D in You
Acronym: STURDY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00063914; U01AG047837 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Vitamin D Deficiency; Falls
Keywords: vitamin D; falls; high risk of falling; insufficient or deficient serum vitamin D levels; 10-29 ng/ml
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 200 IU/d (Active Comparator): 200 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually
  Interventions: Dietary Supplement: 200 IU/d cholecalciferol
- 1000 IU/d (Active Comparator): 1000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually
  Interventions: Dietary Supplement: 1000 IU/d cholecalciferol
- 2000 IU/d (Active Comparator): 2000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually
  Interventions: Dietary Supplement: 2000 IU/d cholecalciferol
- 4000 IU/d (Active Comparator): 4000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually
  Interventions: Dietary Supplement: 4000 IU/d cholecalciferol

INTERVENTIONS:
Dietary Supplement: 200 IU/d cholecalciferol
  Other Names: vitamin D3
  Arms: 200 IU/d
Dietary Supplement: 1000 IU/d cholecalciferol
  Other Names: vitamin D3
  Arms: 1000 IU/d
Dietary Supplement: 2000 IU/d cholecalciferol
  Other Names: vitamin D3
  Arms: 2000 IU/d
Dietary Supplement: 4000 IU/d cholecalciferol
  Other Names: vitamin D3
  Arms: 4000 IU/d

SUMMARY:
Vitamin D supplements might substantially reduce the risk of falls, potentially by more than 25%. The proposed study is a clinical trial that will determine the effects of 4 doses of vitamin D (200 International Units [IU]/day, 1000 IU/day, 2000 IU/d and 4000 IU/d) as a means to prevent falls in high-risk adults, ages 70 and older. Results of this trial will be directly relevant to public health and clinical guidelines, and will immediately influence policy.

DETAILED DESCRIPTION:
The public health burden of falls in older persons is substantial. Several lines of evidence suggest that vitamin D supplements might reduce the risk of falls, potentially by 25% or more in persons with low serum 25-hydroxyvitamin D [25(OH)D] levels. However, existing evidence is inconsistent and insufficient to guide policy. The trial is a seamless two-stage, Bayesian response-adaptive, randomized dose-finding trial designed to select the best dose of vitamin D supplementation and to potentially confirm the efficacy of that dose for fall prevention and other related outcomes. Participants will be community-dwelling adults, aged 70+ (goal of ~40% black, ~60% women), with a baseline serum 25(OH)D level of 10-29 ng/ml, who are at high risk for falling.

In Stage 1 of the adaptive design, participants will be randomly assigned to one of four vitamin D3 (cholecalciferol) doses: 200 IU/d (control), 1000 IU/d, 2000 IU/d, or 4000 IU/d, with assignment probabilities that will vary as falls are reported. Participants will take their assigned pills for two years, or until the study ends, whichever comes first. This stage of the design will select the best non control dose of vitamin D for prevention of falls, or confirm the futility of distinguishing any differences among the non control doses for fall prevention. If a best dose is selected, subsequent participants will be randomized in Stage 2 of the trial into the comparison (200 IU/d) or best dose group, and all participants (Stage 1 and Stage 2) will continue to be followed to potentially confirm efficacy. The investigators anticipate enrolling approximately 1,200 participants over the entire length of the project.

The primary outcome is time to first fall (or death) over two years of therapy. Next in importance is the outcome of gait speed. Other outcomes include fall rates, types of falls, balance, muscle strength, frailty, Short Physical Performance Battery (SPPB) score, 6-minute walk time, and physical activity assessed by accelerometry. Falls will be ascertained from fall calendars completed daily by participants and from self-report by phone. In-person follow-up visits will occur at 3, 12, and 24 months, with telephone visits occurring at 1, 6, 9, 15, 18, and 21 months after randomization. Subgroups with potential for greater benefit from vitamin D supplementation are blacks, those with baseline 25(OH)D of 10-19 ng/ml, and those with objective evidence of low physical function.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 and older
* Non-institutionalized
* High risk for falling, defined by a 'yes' response to at least one of the following:
* 1. Have you fallen and hurt yourself in the past year?
* 2. Have you fallen 2 or more times in the past year?
* 3. Are you afraid that you might fall because of balance or walking problems?
* 4. Do you have difficulty maintaining your balance when bathing, dressing, or getting in and out of a chair?
* 5. Do you use a cane, walker, or other device when walking inside or outside your home?
* Serum vitamin D [25(OH)D] level of 10-29 ng/ml
* Able to provide informed consent
* Willing to accept randomization to each vitamin D dose
* One of the following:
* 1. No vitamin D supplementation at baseline
* 2. Average daily vitamin D supplementation judged by study staff as being consistent with the goal of 1000 IU/day or less at screening and willing to continue the dose unchanged throughout the trial
* One of the following:
* 1. No calcium supplementation at baseline
* 2. Average daily calcium supplementation judged by study staff as being consistent with the goal of 1200 mg/day or less at screening and willing to continue the dose unchanged throughout the trial

Exclusion Criteria:

* Cognitive impairment, defined by Mini-Mental State Exam (MMSE) score <24
* Hypercalcemia, serum Ca++ 11.0 mg/dl or higher or >10.5 mg/dl (confirmed)
* Hypocalcemia, serum Ca++ <8.5 mg/dl
* Kidney, ureteral, or bladder stones made of calcium compounds (2 or more in lifetime, or 1 in the last 2 years); in the absence of information on the type of stone, stones will be assumed to be made of calcium compounds
* Planning to move out of area within 2 years, where plans would prevent compliance with the study protocol
* Disease or condition expected to cause death or to prevent compliance with the study protocol in the next 2 years
* Participation in another trial of vitamin D or falls, or any trial that might affect the risk of falls
* Lactose allergy (lactose intolerance is okay)
* Use of any form of oral or injected calcitriol (brand names: Rocaltrol (R), Calcijex (R), and Zemplar (R); generic names: calcitriol, paricalcitol, doxycalcitriol, 22-oxacalcitriol)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 688 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Appel, MD, MPH, Study Chair — Johns Hopkins University
Locations (2):
- United States (2):
  - ProHealth Clinical Research Unit, Baltimore, Maryland
  - Comstock Center for Public Health Research and Prevention, Hagerstown, Maryland

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data and data dictionary will be available at https://archive.data.jhu.edu/ starting one year after publication of the primary outcome results, contingent upon Institutional Review Board (IRB) approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after publication of primary outcome results. Data are expected to be available in December 2021. Data are expected to remain available in perpetuity.
Access Criteria: Data will be available at https://archive.data.jhu.edu/ contingent on IRB approval of their use.
URL: https://archive.data.jhu.edu/

REFERENCES:
- [Derived] Juraschek SP, Appel LJ, Lipsitz LA, Miller ER 3rd. Reply to: Comment on: Comparison of supine and seated orthostatic hypotension assessments and their association with falls and orthostatic symptoms. J Am Geriatr Soc. 2023 Feb;71(2):674-676. doi: 10.1111/jgs.18113. Epub 2022 Nov 10. No abstract available. PMID 36356235
- [Derived] Michos ED, Kalyani RR, Blackford AL, Sternberg AL, Mitchell CM, Juraschek SP, Schrack JA, Wanigatunga AA, Roth DL, Christenson RH, Miller ER 3rd, Appel LJ. The Relationship of Falls With Achieved 25-Hydroxyvitamin D Levels From Vitamin D Supplementation: The STURDY Trial. J Endocr Soc. 2022 Apr 16;6(6):bvac065. doi: 10.1210/jendso/bvac065. eCollection 2022 Jun 1. PMID 35592513
- [Derived] Juraschek SP, Appel LJ, M Mitchell C, Mukamal KJ, Lipsitz LA, Blackford AL, Cai Y, Guralnik JM, Kalyani RR, Michos ED, Schrack JA, Wanigatunga AA, Miller ER 3rd. Comparison of supine and seated orthostatic hypotension assessments and their association with falls and orthostatic symptoms. J Am Geriatr Soc. 2022 Aug;70(8):2310-2319. doi: 10.1111/jgs.17804. Epub 2022 Apr 22. PMID 35451096
- [Derived] Cai Y, Wanigatunga AA, Mitchell CM, Urbanek JK, Miller ER 3rd, Juraschek SP, Michos ED, Kalyani RR, Roth DL, Appel LJ, Schrack JA. The effects of vitamin D supplementation on frailty in older adults at risk for falls. BMC Geriatr. 2022 Apr 10;22(1):312. doi: 10.1186/s12877-022-02888-w. PMID 35399053
- [Derived] Urbanek JK, Roth DL, Karas M, Wanigatunga AA, Mitchell CM, Juraschek SP, Cai Y, Appel LJ, Schrack JA. Free-Living Gait Cadence Measured by Wearable Accelerometer: A Promising Alternative to Traditional Measures of Mobility for Assessing Fall Risk. J Gerontol A Biol Sci Med Sci. 2023 May 11;78(5):802-810. doi: 10.1093/gerona/glac013. PMID 35029661
- [Derived] Guralnik JM, Sternberg AL, Mitchell CM, Blackford AL, Schrack J, Wanigatunga AA, Michos E, Juraschek SP, Szanton S, Kalyani R, Cai Y, Appel LJ; STURDY Collaborative Research Group. Effects of Vitamin D on Physical Function: Results From the STURDY Trial. J Gerontol A Biol Sci Med Sci. 2022 Aug 12;77(8):1585-1592. doi: 10.1093/gerona/glab379. PMID 34928336
- [Derived] Miller HN, Plante TB, Gleason KT, Charleston J, Mitchell CM, Miller ER 3rd, Appel LJ, Juraschek SP. A/B design testing of a clinical trial recruitment website: A pilot study to enhance the enrollment of older adults. Contemp Clin Trials. 2021 Dec;111:106598. doi: 10.1016/j.cct.2021.106598. Epub 2021 Oct 12. PMID 34653651
- [Derived] Juraschek SP, Miller ER, Wanigatunga AA, Schrack JA, Michos ED, Mitchell CM, Kalyani RR, Appel LJ. Effects of Vitamin D Supplementation on Orthostatic Hypotension: Results From the STURDY Trial. Am J Hypertens. 2022 Feb 1;35(2):192-199. doi: 10.1093/ajh/hpab147. PMID 34537827
- [Derived] Appel LJ, Michos ED, Mitchell CM, Blackford AL, Sternberg AL, Miller ER 3rd, Juraschek SP, Schrack JA, Szanton SL, Charleston J, Minotti M, Baksh SN, Christenson RH, Coresh J, Drye LT, Guralnik JM, Kalyani RR, Plante TB, Shade DM, Roth DL, Tonascia J; STURDY Collaborative Research Group. The Effects of Four Doses of Vitamin D Supplements on Falls in Older Adults : A Response-Adaptive, Randomized Clinical Trial. Ann Intern Med. 2021 Feb;174(2):145-156. doi: 10.7326/M20-3812. Epub 2020 Dec 8. PMID 33284677
- [Derived] Plante TB, Gleason KT, Miller HN, Charleston J, McArthur K, Himmelfarb CD, Lazo M, Ford DE, Miller ER 3rd, Appel LJ, Juraschek SP; STURDY Collaborative Research Group. Recruitment of trial participants through electronic medical record patient portal messaging: A pilot study. Clin Trials. 2020 Feb;17(1):30-38. doi: 10.1177/1740774519873657. Epub 2019 Oct 3. PMID 31581836
- [Derived] Michos ED, Mitchell CM, Miller ER 3rd, Sternberg AL, Juraschek SP, Schrack JA, Szanton SL, Walston JD, Kalyani RR, Plante TB, Christenson RH, Shade D, Tonascia J, Roth DL, Appel LJ; STURDY Collaborative Research Group. Rationale and design of the Study To Understand Fall Reduction and Vitamin D in You (STURDY): A randomized clinical trial of Vitamin D supplement doses for the prevention of falls in older adults. Contemp Clin Trials. 2018 Oct;73:111-122. doi: 10.1016/j.cct.2018.08.004. Epub 2018 Aug 20. PMID 30138718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2015 to March 2018, new participants were randomized in the trial's Stage 1 and began their individual 2-year period of trial participation. Stage 1 ended on March 23, 2018 and Stage 2 began; randomization continued but to the 200 and 1000 groups only. Some participants completed their 2 years of participation during Stage 1, some participants had follow-up time during both Stage 1 and Stage 2, and some participants began their 2 years of participation during Stage 2.
Groups:
- Randomized to 200 IU/d in Stage 1: These participants received 200 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually throughout their trial participation; those who continued to Stage 2 (neither completed the trial [completed the 2-year visit], nor died, nor dropped out during Stage 1) continued to receive 200 IU/d cholecalciferol during Stage 2.
- Additional Participants Randomized to 200 IU/d in Stage 2: These participants began their study participation in Stage 2 and received 200 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually throughout their participation.
- Randomized to 1000 IU/d in Stage 1: These participants received 1000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually throughout their trial participation; those who continued to Stage 2 (neither completed the trial [completed the 2-year visit], nor died, nor dropped out during Stage 1) continued to receive 1000 IU/d cholecalciferol during Stage 2.
- Additional Participants Randomized to 1000 IU/d in Stage 2: These participants began their study participation in Stage 2 and received 1000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually throughout their participation.
- Randomized to 2000 IU/d in Stage 1 and Switched to 1000 IU/d in Stage 2: These participants received 2000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually in Stage 1; those who continued to Stage 2 were switched to 1000 IU/d cholecalciferol (vitamin D3) tablets during Stage 2.
- Randomized to 4000 IU/d in Stage 1 and Switched to 1000 IU/d in Stage 2: These participants received 4000 IU/d cholecalciferol (vitamin D3) tablets that can be swallowed or consumed sublingually in Stage 1; those who continued to Stage 2 were switched to 1000 IU/d cholecalciferol (vitamin D3) tablets during Stage 2.
Period: Stage 1
Arm/Group | Randomized to 200 IU/d in Stage 1 | Additional Participants Randomized to 200 IU/d in Stage 2 | Randomized to 1000 IU/d in Stage 1 | Additional Participants Randomized to 1000 IU/d in Stage 2 | Randomized to 2000 IU/d in Stage 1 and Switched to 1000 IU/d in Stage 2 | Randomized to 4000 IU/d in Stage 1 and Switched to 1000 IU/d in Stage 2
Started | 262 | 0 | 130 | 0 | 68 (Randomization to 2000 IU/d was stopped in February 2018 as part of planned dose-finding) | 69 (Randomization to 4000 IU/d was stopped in March 2018 as part of planned dose-finding)
Completed (In Stage 1, completed = started Stage 2) | 242 | 0 | 122 | 0 | 59 | 63
Not Completed | 20 | 0 | 8 | 0 | 9 | 6
Not completed — Finished the trial (did the 2 year visit) during Stage 1 and did not advance to Stage 2 | 4 | 0 | 0 | 0 | 3 | 1
Not completed — Death | 4 | 0 | 2 | 0 | 3 | 2
Not completed — Lost to Follow-up | 12 | 0 | 6 | 0 | 3 | 3
Period: Stage 2
Arm/Group | Randomized to 200 IU/d in Stage 1 | Additional Participants Randomized to 200 IU/d in Stage 2 | Randomized to 1000 IU/d in Stage 1 | Additional Participants Randomized to 1000 IU/d in Stage 2 | Randomized to 2000 IU/d in Stage 1 and Switched to 1000 IU/d in Stage 2 | Randomized to 4000 IU/d in Stage 1 and Switched to 1000 IU/d in Stage 2
Started | 242 | 77 | 122 | 82 | 59 | 63
Completed (In Stage 2, completed = participated in closeout (April-May 2019)) | 35 | 71 | 47 | 73 | 2 | 4
Not Completed | 207 | 6 | 75 | 9 | 57 | 59
Not completed — Finished the trial (did the 2 year visit) prior to or during trial closeout | 180 | 0 | 63 | 0 | 54 | 52
Not completed — Death | 4 | 2 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 23 | 4 | 11 | 9 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- 200 IU/d: The 200 IU/d group is the control group.
- 1000 IU/d: During dose-finding, the 1000 IU/d dose was identified as the best of the non-control doses for fall prevention.
- 2000 IU/d: Randomization to the 2000 IU/d group was stopped in February 2018 as part of planned dose-finding.
- 4000 IU/d: Randomization to the 4000 IU/d group was stopped in March 2018 as part of planned dose-finding.
- Total: Total of all reporting groups
Arm/Group | 200 IU/d | 1000 IU/d | 2000 IU/d | 4000 IU/d | Total
Number analyzed (Participants) | 339 | 212 | 68 | 69 | 688
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (5.4) | 76.5 (5.3) | 77.3 (4.6) | 79.1 (5.9) | 77.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 102 | 29 | 28 | 300
  Male | 198 | 110 | 39 | 41 | 388
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 7 participants were missing race information, 4 participants were missing ethnicity information
  Participants
    White: number analyzed (Participants) | 335 | 210 | 67 | 69 | 681
    White | 276 | 159 | 51 | 57 | 543
    Black: number analyzed (Participants) | 335 | 210 | 67 | 69 | 681
    Black | 55 | 44 | 15 | 10 | 124
    Other: number analyzed (Participants) | 335 | 210 | 67 | 69 | 681
    Other | 7 | 12 | 2 | 2 | 23
    Hispanic, Latino or Spanish ethnicity: number analyzed (Participants) | 336 | 211 | 68 | 69 | 684
    Hispanic, Latino or Spanish ethnicity | 3 | 3 | 1 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 339 | 212 | 68 | 69 | 688
Serum vitamin D (nmol/L) [Count of Participants; unit: Participants] — The range of serum vitamin D levels eligible for the trial (25-72.5 nmol/L) includes those termed deficient (<50 nmol/L) or insufficient (50-72.5 nmol/L) by the Endocrine Society and overlaps with those termed deficient (<30 nmol/L), inadequate (30 to <50 nmol/L), or adequate (≥50 nmol/L) by the Institute of Medicine.
  Participants
    25 to 49 nmol/L | 100 | 53 | 25 | 22 | 200
    50 to 72.5 nmol/L | 239 | 159 | 43 | 47 | 488
Taking a vitamin D supplement [Count of Participants; unit: Participants] | 124 | 82 | 27 | 23 | 256
Total vitamin D intake (IU/day) [Count of Participants; unit: Participants]
  < 200 | 125 | 77 | 21 | 30 | 253
  200-399 | 68 | 40 | 16 | 14 | 138
  400-799 | 63 | 39 | 10 | 13 | 125
  >= 800 | 83 | 56 | 21 | 12 | 172
Fell at least once in prior year [Count of Participants; unit: Participants] | 221 | 139 | 43 | 47 | 450
Fell and hurt self in prior year [Count of Participants; unit: Participants] | 130 | 81 | 21 | 30 | 262
Fell at least twice in prior year [Count of Participants; unit: Participants] | 120 | 83 | 26 | 30 | 259
Afraid of falling due to balance or walking problem [Count of Participants; unit: Participants] — Population: 1 participant in the 1000 IU/day group did not answer the question regarding fear of falling due to balance or walking problem.
  Participants
    number analyzed (Participants) | 339 | 211 | 68 | 69 | 687
    (all) | 290 | 190 | 65 | 56 | 601
Difficulty maintaining balance [Count of Participants; unit: Participants] | 173 | 99 | 33 | 38 | 343
Uses cane, walker or other assistive device to walk [Count of Participants; unit: Participants] — Population: 1 participant in the 1000 IU/day group did not answer the question about using an assistive device to walk.
  Participants
    number analyzed (Participants) | 339 | 211 | 68 | 69 | 687
    (all) | 91 | 64 | 24 | 25 | 204
Short Physical Performance Battery score [Count of Participants; unit: Participants] — The Short Physical Performance Battery (SPPB) is a 3-part assessment of physical functioning: balance testing, gait speed testing (timed 4-meter walk at usual pace), and demonstration of ability to complete 5 chair stands; each part is scored 0 to 4 and the 3 subscores are summed to obtain the total score which ranges from 0 to 12. Higher scores indicate better physical function.
  Participants
    0 to 3 | 12 | 12 | 3 | 3 | 30
    4 to 6 | 34 | 18 | 12 | 11 | 75
    7 to 9 | 131 | 92 | 30 | 24 | 277
    10 to 12 | 162 | 90 | 23 | 31 | 306
Gait speed (m/sec) [Mean (Standard Deviation); unit: meters per second] — Population: 1 participant in the 200 IU/day group and 2 participants in the 1000 IU/day group were missing gait speed at baseline
  meters per second
    number analyzed (Participants) | 338 | 210 | 68 | 69 | 685
    (all) | 0.89 (0.23) | 0.85 (0.23) | 0.80 (0.23) | 0.85 (0.23) | 0.86 (0.24)
Frailty status [Count of Participants; unit: Participants] — Population: One participant in the 1000 IU/day group was missing frailty status at baseline.
  Participants
    number analyzed (Participants) | 339 | 211 | 68 | 69 | 687
    Robust | 104 | 51 | 25 | 18 | 198
    Pre-frail | 205 | 127 | 36 | 40 | 408
    Frail | 30 | 33 | 7 | 11 | 81
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: 1 participant in the 1000 IU/day group was missing BMI at baseline.
  kg/m^2
    number analyzed (Participants) | 339 | 211 | 68 | 69 | 687
    (all) | 30.4 (6.3) | 30.7 (5.2) | 30.7 (6.4) | 30.3 (6.2) | 30.5 (6.0)
SF-12 physical health component score [Mean (Standard Deviation); unit: units on a scale] — The Short-Form 12-Item Health Survey (4-week recall) v2 (SF-12) is an interviewer-administered 12-item scale measuring a person's perceptions of their health and health-related quality of life; the physical component score is based on responses to 6 items and has a normative mean (SD) of 50 (10) (range 0 to 100). Higher scores indicate better physical health. Population: 4 participants in the 200 IU/day group and 1 participant in the 1000 IU/day group were missing the SF-12 physical component score at baseline.
  units on a scale
    number analyzed (Participants) | 335 | 211 | 68 | 69 | 683
    (all) | 44.5 (10.3) | 42.9 (11.0) | 42.9 (10.2) | 44.0 (9.9) | 43.8 (10.5)
SF-12 mental health component score [Mean (Standard Deviation); unit: units on a scale] — The Short-Form 12-Item Health Survey (4-week recall) v2 (SF-12) is an interviewer-administered 12-item scale measuring a person's perceptions of their health and health-related quality of life; the mental component score is based on responses to 6 items and has a normative mean (SD) of 50 (10) (range 0 to 100). Higher scores indicate better mental health. Population: 4 participants in the 200 IU/day group and 1 participant in the 1000 IU/day group were missing the SF-12 mental component score at baseline.
  units on a scale
    number analyzed (Participants) | 335 | 211 | 68 | 69 | 683
    (all) | 55.1 (7.7) | 55.4 (7.6) | 54.5 (8.4) | 54.3 (9.4) | 55.0 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of First Fall or Death (Whichever Comes First)
Description: Falls were ascertained by a monthly fall calendar completed by each participant, scheduled interviews at 1 month and 3 months after randomization and every 3 months thereafter up to 24 months or trial end. Death was ascertained primarily by reports from family or friends.
Time Frame: Randomization to 24 months or end of trial, whichever came first
Population: The primary efficacy analysis compares the Experience on Best Dose group versus the 200 IU/d group. The Experience on Best Dose group includes all participants assigned or switched to best dose, with their data limited to data while on best dose. This group excludes 41 participants randomized to 2000 or 4000 IU/d who were never issued a bottle of 1000 IU/d because they completed the trial, died, dropped out, or stopped using study pills without ever being switched to 1000 IU/d.
Measure: Number (95% Confidence Interval); unit: First fall or death per 100 person-years
Groups:
- Experience on Best Dose: The Experience on Best Dose group includes 121 participants randomized to 1000 IU/d during dose-finding and 96 participants randomized to 2000 or 4000 IU/d during dose-finding who were issued at least one bottle of 1000 IU after dose-finding ended, plus 91 participants randomized to 1000 IU/d after dose-finding ended, for a total of 308 participants who had experience on the dose selected as best of the non-control doses for preventing falls. This group excludes 41 participants randomized to 2000 or 4000 IU/d who were never issued a bottle of 1000 IU/d because they completed the trial, died, dropped out, or stopped using study pills without ever being switched to 1000 IU/d.
- 200 IU/d: The 200 IU/d group is the control group and includes participants randomized to 200 IU/d during Stage 1 and participants randomized to 200 IU/d during Stage 2.
- Pooled Higher Doses: All participants randomized to 1000, 2000, or 4000 IU/d during Stage 1 and all participants randomized to 1000 IU/d during Stage 2.
Arm/Group | Experience on Best Dose | 200 IU/d | Pooled Higher Doses
Number analyzed (Participants) | 308 | 339 | 349
First fall or death per 100 person-years | 76.9 [65.8 to 89.9] | 76.0 [66.5 to 86.9] | 78.0 [68.3 to 89.0]
Statistical Analysis 1: Comparison: Experience on Best Dose vs 200 IU/d; The Experience on Best Dose group includes all participants assigned or switched to best dose (1000 IU/day) and excludes 41 participants randomized to 2000 or 4000 IU/day who were never issued a bottle of best dose. For those randomized to 2000 or 4000 IU/day, at-risk time and events are measured from the date of their switch to best dose. 150 Experience on Best Dose participants (median follow-up, 10.2 mos) and 125 200 IU/day participants (median follow-up, 20.3 mos) were censored; Test type: Superiority; p = 0.54, Log Rank — The P value is nominal and two-sided; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.76 to 1.15] — The Experience on Best Dose versus 200 IU/day hazard ratio and its 95% confidence interval were derived from a Cox regression model with dose group as the single model variable
Statistical Analysis 2: Comparison: 200 IU/d vs Pooled Higher Doses; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.86 to 1.25] — The comparison of the Pooled Higher Doses group versus the 200 IU/d group is a sensitivity analysis

2. Secondary Outcome: Change in Gait Speed
Description: Gait speed in meters per second (m/s) was obtained from the timed 4-meter, usual-paced walk component of the Short Physical Performance Battery. The change in gait speed was obtained as follow-up measure minus baseline measure.
Time Frame: Baseline, 3 months, 12 months and 24 months
Population: Change in gait speed since randomization was evaluated in the Pooled Higher Doses group versus the 200 IU/d group.
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Pooled Higher Doses: The Pooled Higher Doses group includes all participants randomized to 1000, 2000, or 4000 IU/d (n=349).
- 200 IU/Day: The 200 IU/d group is the control group.
Arm/Group | Pooled Higher Doses | 200 IU/Day
Number analyzed (Participants) | 349 | 339
m/s
  Change at 3 months | -0.01 (0.17) | -0.01 (0.18)
  Change at 12 months | -0.04 (0.17) | -0.04 (0.20)
  Change at 24 months | -0.03 (0.16) | -0.09 (0.21)
Statistical Analysis 1: Comparison: Pooled Higher Doses vs 200 IU/Day; The two groups were assessed for differential change over time in change from baseline using a longitudinal mixed effects regression model with gait speed as the outcome and fixed effects including a single treatment term, 3 time point terms and 3 treatment-by-time interaction terms and a random intercept for participant; Test type: Superiority — The overall P tests for difference between groups in differential change from baseline over time and is from a 3 degree of freedom test of the combined 3 treatment-by-time interaction terms from the longitudinal mixed effects model; p = 0.15, Regression, Linear — The P value is nominal and not adjusted for multiple comparisons; 3 degree of freedom interaction test

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from randomization to last date of participation in the trial, up to 24 months.
Description: Adverse events are reported for the Pooled Higher Doses group (those randomized to 1000, 2000, or 4000 IU) vs. the control group (those randomized to 200 IU) to be consistent with how the study outcomes are reported, because the Pooled Higher Doses and control groups have comparable numbers and follow-up, and because the 2000 and 4000 IU groups received 1000 IU after 1000 IU was selected as best non control dose. Also shown are counts of adverse event by dose in use when the event occurred.
Groups:
- Pooled Higher Doses: The Pooled Higher Doses group includes all participants randomized to 1000, 2000, or 4000 IU/d.
- Those With Experience on 1000 IU: This group includes those randomized to 1000 IU and 96 participants randomized to 2000 or 4000 who were issued at least 1 bottle of 1000 IU. Note that participants who switched doses during the trial may have an event while in their original group as well as in the 1000 group if the event recurred after switching to 1000 IU.
- Those With Experience on 2000 IU: Only those randomized to 2000 IU are in this group.
- Those With Experience on 4000 IU: Only those randomized to 4000 IU are in this group.
Arm/Group | Pooled Higher Doses | 200 IU/d | Those With Experience on 1000 IU | Those With Experience on 2000 IU | Those With Experience on 4000 IU
All-Cause Mortality (participants affected / at risk) | 9/349 | 10/339 | 4/308 | 3/68 | 2/69
Serious Adverse Events (participants affected / at risk) | 82/349 | 68/339 | 49/308 | 17/68 | 17/69
Other Adverse Events (participants affected / at risk) | 311/349 | 299/339 | 250/308 | 60/68 | 63/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Higher Doses (N=349) | 200 IU/d (N=339) | Those With Experience on 1000 IU (N=308) | Those With Experience on 2000 IU (N=68) | Those With Experience on 4000 IU (N=69)
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 2 | 0
Cardiac disorder (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 3 | 1 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Gastrointestinal polyp hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 3 | 1 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 0
Abasia (General disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 2 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Medical device complication (General disorders) | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 1 | 0
Polyp (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1 | 0 | 1
Unevaluable event (General disorders) | 1 | 1 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 3 | 1 | 1 | 0
Localized infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 6 | 2 | 4 | 1
Sepsis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 | 1 | 1
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 1 | 4 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 1
Full blood count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung cancer metastatis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 3 | 2 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0 | 1
Hemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Dypsnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 2 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 1 | 0 | 0
Internal hemorrhage (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 3 | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Fecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Device malfunction (General disorders) | 1 | 0 | 0 | 0 | 1
Necrosis (General disorders) | 1 | 0 | 1 | 0 | 0
Ulcer (General disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 1 | 1 | 1 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Prostatic calcification (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Higher Doses (N=349) | 200 IU/d (N=339) | Those With Experience on 1000 IU (N=308) | Those With Experience on 2000 IU (N=68) | Those With Experience on 4000 IU (N=69)
Diarrhea (Gastrointestinal disorders) | 26 | 19 | 16 | 4 | 6
Nausea (Gastrointestinal disorders) | 65 | 57 | 44 | 9 | 13
Vomiting (Gastrointestinal disorders) | 38 | 31 | 25 | 7 | 7
Contusion (Injury, poisoning and procedural complications) | 112 | 92 | 71 | 23 | 24
Influenza (Infections and infestations) | 14 | 17 | 9 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 212 | 207 | 153 | 44 | 47
Ligament sprain (Injury, poisoning and procedural complications) | 20 | 15 | 14 | 2 | 4
Muscle strain (Injury, poisoning and procedural complications) | 58 | 49 | 37 | 5 | 18
Skin abrasion (Injury, poisoning and procedural complications) | 95 | 85 | 54 | 22 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 34 | 20 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 26 | 22 | 18 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 14 | 14 | 4 | 4
Dizziness (Nervous system disorders) | 26 | 25 | 18 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02166333/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT02166333/SAP_001.pdf